CLINICAL TRIAL: NCT06779708
Title: ECHO-NET Study: Role of Intraoperative Hepatic Ultrasonography in Patients with Gastrointestinal or Pancreatic Neuroendocrine Tumor Without Liver Metastases At Preoperative Imaging
Brief Title: The Role of Intraoperative Hepatic Ultrasonography in Gastrointestinal or Pancreatic Neuroendocrine Tumor
Acronym: ECHO-NET
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 748/2020
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine (NE) Tumors; Liver Metastasis
Keywords: neuroendocrine tumors; liver metastases; intraoperative hepatic ultrasonography
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Liver metastases are common in patients with neuroendocrine neoplasms, but often underestimated by preoperative imaging. Intraoperative ultrasound (IOUS) is the reference standard for staging of primary and metastatic liver tumors, with a diagnostic accuracy superior to that of CT and MRI. Rationale: The present study aims to evaluate the contribution of IOUS to staging of liver disease in patients with neuroendocrine tumor candidates for primary tumor resection classified as cM0 at preoperative imaging.

The study will collect a prospective series of 99 patients undegoing surgery for gastro-intestinal or pancreatic neuroendocrine tumor at the Humanitas Clinical Institute (coordinating centre) or at one of the participating centres in the period 2020-2023. All patients had to be cM0 tumor at preoperative imaging. Additional inclusion criteria: age>18 years, ability to give the informed consent for study participation; no other malignancies in the previous 5 years; preoperative staging including abdominal CT and DOTATOC PET-CT performed ≤60 days before surgery.

This prospective observational multicentre study aims to elucidate the proportion of patients with gastro-intestinal or pancreatic neuroendocrine tumor cM0 at preoperative imaging that have intraoperative detection of liver metastases at IOUS.

Primary endpoint:

- Performances of IOUS in identifying liver metastases in patients with neuroendocrine tumor classified as cM0 at preoperative imaging

Secondary endpoints:

* Impact of IOUS on the therapeutic strategy
* Performances of preoperative imaging (CT, MRI and PET-CT) in comparison with those of IOUS

The study will collect a prospective series of 99 patients undergoing surgery for gastro-intestinal or pancreatic neuroendocrine tumor at the Humanitas Clinical Institute (coordinating centre) or at one of the participating centres in the period 2020-2023.

The study includes the following steps:

Preoperative / enrollment: All patients candidates to resection of gastro-intestinal or pancreatic neuroendocrine tumor will be considered for the study. Only cM0 patients will be enrolled. All patients enrolled in the study must have performed a preoperative abdominal CT scan with contrast medium and a DOTATOC-PET-CT (both performed ≤60 days before surgery).

Intraoperative: During surgery, the investigator will perform, as standard in our clinical practice, an accurate exploration of the liver by inspection, palpation and IOUS. The investigator will record the identification of any liver lesion. If one or more nodules suspect of being neuroendocrine liver metastases are identified, it will be necessary, whenever possible, as already routinely performed, to carry out a biopsy or to remove it (if superficial) for histological confirmation of the diagnosis. After completion of liver staging, the primary tumor will be resected.

Postoperative / follow-up: Enrolled patients will have standard postoperative management.

Standard statistical analyses will be performed. Per-patient and per-lesion analyses will be performed to asses performances of preoperative imaging modalities (CT, MRI, PET-CT) and of intraoperative ones (inspection, palpation, and IOUS).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open or minimally-invasive surgery for primary neuroendocrine gastro-intestinal or pancreatic tumor.
* cM0 tumor at preoperative imaging
* Preoperative staging including abdominal CT and DOTATOC PET-CT
* Age ≥18 years
* No other malignancies in the previous 5 years

Exclusion Criteria:

* Preoperative imaging performed >60 days before surgery
* Patient refusal to participate the study
* Incomplete intraoperative hepatic staging (peri-hepatic adhesions, IOUs not available…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will collect a prospective series of 99 patients undergoing surgery for gastro-intestinal or pancreatic neuroendocrine tumor at the Humanitas Clinical Institute (coordinating centre) or at one of the participating centres (see the Appendix for list of the centres) in the period 2020-2023.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Liver metastases | 2020-2023
  Performances of IOUS in identifying liver metastases in patients with neuroendocrine tumor classified as cM0 at preoperative imaging

SECONDARY OUTCOMES:
Impact on therapeutic strategies | 2020-2023
Comparison with radiological preoperative evaluation | 2020-2023
  Performances of preoperative imaging (CT, MRI and PET-CT) in comparison with those of IOUS

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vigano L, Ferrero A, Amisano M, Russolillo N, Capussotti L. Comparison of laparoscopic and open intraoperative ultrasonography for staging liver tumours. Br J Surg. 2013 Mar;100(4):535-42. doi: 10.1002/bjs.9025. Epub 2013 Jan 21. PMID 23339035
- [Background] Langella S, Ardito F, Russolillo N, Panettieri E, Perotti S, Mele C, Giuliante F, Ferrero A. Intraoperative Ultrasound Staging for Colorectal Liver Metastases in the Era of Liver-Specific Magnetic Resonance Imaging: Is It Still Worthwhile? J Oncol. 2019 Sep 22;2019:1369274. doi: 10.1155/2019/1369274. eCollection 2019. PMID 31662749
- [Background] Torzilli G, Botea F, Donadon M, Cimino M, Procopio F, Pedicini V, Poretti D, Montorsi M. Criteria for the selective use of contrast-enhanced intra-operative ultrasound during surgery for colorectal liver metastases. HPB (Oxford). 2014 Nov;16(11):994-1001. doi: 10.1111/hpb.12272. Epub 2014 May 15. PMID 24830573
- [Background] van Vledder MG, Pawlik TM, Munireddy S, Hamper U, de Jong MC, Choti MA. Factors determining the sensitivity of intraoperative ultrasonography in detecting colorectal liver metastases in the modern era. Ann Surg Oncol. 2010 Oct;17(10):2756-63. doi: 10.1245/s10434-010-1108-y. Epub 2010 Jun 2. PMID 20517682
- [Background] Elias D, Lefevre JH, Duvillard P, Goere D, Dromain C, Dumont F, Baudin E. Hepatic metastases from neuroendocrine tumors with a "thin slice" pathological examination: they are many more than you think.. Ann Surg. 2010 Feb;251(2):307-10. doi: 10.1097/SLA.0b013e3181bdf8cf. PMID 20010089
- [Background] Ruzzenente A, Bagante F, Bertuzzo F, Aldrighetti L, Campagnaro T, Ercolani G, Conci S, Giuliante F, Dore A, Ferrero A, Torzilli G, Grazi GL, Ratti F, Cucchetti A, De Rose AM, Russolillo N, Cimino M, Perri P, Guglielmi A, Iacono C. Liver Resection for Neuroendocrine Tumor Liver Metastases Within Milan Criteria for Liver Transplantation. J Gastrointest Surg. 2019 Jan;23(1):93-100. doi: 10.1007/s11605-018-3973-9. Epub 2018 Sep 21. PMID 30242647
- [Background] O'Toole D, Kianmanesh R, Caplin M. ENETS 2016 Consensus Guidelines for the Management of Patients with Digestive Neuroendocrine Tumors: An Update. Neuroendocrinology. 2016;103(2):117-8. doi: 10.1159/000443169. Epub 2016 Jan 6. No abstract available. PMID 26731186
- [Background] Hallet J, Law CH, Cukier M, Saskin R, Liu N, Singh S. Exploring the rising incidence of neuroendocrine tumors: a population-based analysis of epidemiology, metastatic presentation, and outcomes. Cancer. 2015 Feb 15;121(4):589-97. doi: 10.1002/cncr.29099. Epub 2014 Oct 13. PMID 25312765
- [Background] Frilling A, Modlin IM, Kidd M, Russell C, Breitenstein S, Salem R, Kwekkeboom D, Lau WY, Klersy C, Vilgrain V, Davidson B, Siegler M, Caplin M, Solcia E, Schilsky R; Working Group on Neuroendocrine Liver Metastases. Recommendations for management of patients with neuroendocrine liver metastases. Lancet Oncol. 2014 Jan;15(1):e8-21. doi: 10.1016/S1470-2045(13)70362-0. PMID 24384494